CLINICAL TRIAL: NCT06993350
Title: Impact of a Targeted 8-Week Exercise Program on Pain Measures and Isokinetic Muscle Strength in Females With Patellofemoral Pain Syndrome: A Randomized Controlled Trial
Brief Title: Impact of a Targeted 8-Week Exercise Program on Pain Measures and Isokinetic Muscle Strength in Females With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Azza Mohammed, Prof. Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Faculty of Physical Therapy; faculty of physical therapy (Registry Identifier: faculty of physical therapy)
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral pain syndrome; weight-bearing pain; isokinetic strength
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (patients with PFPS) (Other): patients receive specific weight bearing program known as weight bearing exercise for better balance program
  Interventions: Other: experimental group
- control group (No Intervention): patient will not receive any intervention

INTERVENTIONS:
Other: experimental group — eight weeks of targeted weight bearing program
  Other Names: weight bearing program
  Arms: group A (patients with PFPS)

SUMMARY:
Patellofemoral pain syndrome (PFPS) is condition characterized by anterior knee pain that predominantly affects young and physically active females. The etiology of PFPS is multifactorial, involving biomechanical, muscular, and neuromuscular factors that contribute to altered patellar tracking and increased pain sensitivity.

DETAILED DESCRIPTION:
This study will employ a randomized controlled trial (RCT) design to evaluate the effects of a targeted 8-week exercise program on pain measures and isokinetic muscle strength in females with PFPS. Thirty female patients diagnosed with PFPS will be recruited based on predefined inclusion and exclusion criteria. Participants will be randomly assigned into two groups: an intervention group receiving the targeted exercise program, and a control group will not receive any intervention.The intervention group will undergo a supervised, structured exercise program lasting 8 weeks, focusing on strengthening the hip and knee muscles, improving neuromuscular control, and addressing pain sensitivity. Sessions will be conducted multiple times per week under professional supervision. Outcome measures will include pain measures, assessed through validated tools such as pressure pain threshold and pain intensity measured by VAS scale and isokinetic muscle strength of knee and hip muscles, measured by isokinetic dynamometry at the Biodex isokinetic Laboratory at the Faculty of Physical Therapy, Cairo University.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will present with clinically diagnosed anterior knee pain exacerbated by activities such as stair climbing, squatting, or prolonged sitting, with a pain duration of at least three months to ensure chronicity. All participants will possess adequate intellectual and cognitive abilities to comprehend and follow exercise instructions, and they will provide informed consent prior to enrollment.

Exclusion Criteria:

Exclusion criteria will include any history of knee surgery or trauma within the past year, presence of other knee pathologies such as ligament injuries or osteoarthritis, neurological or systemic disorders affecting lower limb function, pregnancy, contraindications to exercise, or current involvement in other physical therapy or structured exercise programs targeting the knee.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-02 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
pain intensity | two times of testing (before and 8 weeks after intervention)
  measured by Visual Analogue Scale. a score range from 0 to 10. 0 means no pain and 10 means severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided